CLINICAL TRIAL: NCT01236664
Title: An Evaluation of the Memory at Work Program
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor is no longer developing this program and therefore has withdrawn the funding.
Sponsor: Baycrest (Other)
Collaborators: Cogniciti Inc. (Industry)
Responsible Party: Angela Troyer, Ph.D., Baycrest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB1043; HTX 10-43 (Other Grant/Funding Number: HTX)
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Cognition - Other; Ageing
Keywords: memory training; mnemonics; cognition; work
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memory Training (Experimental)
  Interventions: Behavioral: Memory training
- Control workshop (Active Comparator)
  Interventions: Behavioral: Control Workshop

INTERVENTIONS:
Behavioral: Memory training — The Memory at Work program is a 4-hour classroom-based workshop that is led by a professional trainer. The format of the program is experiential, with a heavy focus on discussion, self-discovery, and hands-on use of trained skills. Specific memory compensation techniques are trained. Training consists of an explanation of each technique (i.e., how and when to use it, the science behind the technique) and ample opportunities for hands-on use of the strategies.
  Other Names: Memory at Work Program
  Arms: Memory Training
Behavioral: Control Workshop — The control workshop consists of a 4-hour program that will train techniques for successfully completing Sudoku, word, and logic puzzles. Like the experimental intervention, the control workshop will be engaging and challenging, and will involve a combination of individual and group activities.
  Arms: Control workshop

SUMMARY:
With the aging of the Canadian population, older workers are accounting for more and more of the working-age population. Despite recent interest in cognitive training, there are currently no validated programs that specifically target individuals in the work force. The investigators will conduct a small-scale randomized controlled trial to test the effectiveness of the previously developed Memory at Work program. The investigators will recruit 60 individuals and randomly assign them to the active intervention or a control intervention. The investigators will examine outcomes related to knowledge, behavioral change, self-efficacy, objective memory, and workplace productivity. The investigators expect larger improvements on these measures in the active relative to the control group.

DETAILED DESCRIPTION:
This is a pre-test/post-test randomized controlled trial. Participants who meet eligibility criteria will undergo baseline testing that involves completing questionnaires and objective cognitive tests. Participants will then be randomly assigned (by coin toss) to the intervention or control group. After participating in their respective workshops, both groups will undergo immediate post-testing and 1-month follow-up post testing. After the final assessment, the control group will be given the opportunity to participate in the intervention workshop. No further testing of this group will occur, as there will no longer be a comparable control group.

ELIGIBILITY:
Inclusion Criteria:

* Currently employed
* Between ages 30-65
* Fluent in English language

Exclusion Criteria:

* A severe head injury, epilepsy or other neurological disorder
* Currently unemployed
* Evidence of significant psychiatric disorder/use of psychotropic medications
* Evidence of substance abuse

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Memory related knowledge and behaviour | 6 weeks

SECONDARY OUTCOMES:
Improved workplace productivity | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Angela K. Troyer, PhD, Principal Investigator — Baycrest; Kelly J Murphy, PhD, Principal Investigator — Baycrest
Locations (1):
- Baycrest, Toronto, Ontario, Canada

REFERENCES:
- [Background] Troyer AK, Murphy KJ, Anderson ND, Moscovitch M, Craik FI. Changing everyday memory behaviour in amnestic mild cognitive impairment: a randomised controlled trial. Neuropsychol Rehabil. 2008 Jan;18(1):65-88. doi: 10.1080/09602010701409684. PMID 17943615
- [Background] Troyer AK, Hafliger A, Cadieux MJ, Craik FI. Name and face learning in older adults: effects of level of processing, self-generation, and intention to learn. J Gerontol B Psychol Sci Soc Sci. 2006 Mar;61(2):P67-74. doi: 10.1093/geronb/61.2.p67. PMID 16497956
- [Background] Troyer AK, Rich JB. Psychometric properties of a new metamemory questionnaire for older adults. J Gerontol B Psychol Sci Soc Sci. 2002 Jan;57(1):P19-27. doi: 10.1093/geronb/57.1.p19. PMID 11773220
- [Background] Troyer AK. Improving memory knowledge, satisfaction, and functioning via an education and intervention program for older adults. Aging, Neuropsychology, and Cognition 8, 256-268, 2001.